CLINICAL TRIAL: NCT06961357
Title: Phase I/II Clinical Trial of CD40L-augmented Tumor Infiltrating Lymphocytes (TIL) for Patients With Advanced Melanoma
Brief Title: Clinical Trial of CD40L-augmented TIL for Patients With Advanced Melanoma
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: MCC-23082
Record Dates: First submitted 2025-04-29; First posted 2025-05-07 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-12

CONDITIONS: Melanoma
Keywords: Mucosal melanoma; Uveal melanoma; Cutaneous acral melanoma; Cutaneous non-acral melanoma
MeSH Terms: conditions — Melanoma; Uveal Melanoma | interventions — Cyclophosphamide; fludarabine; Interleukin-2

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Cohort 1: Phase I safety trial (Experimental): Participants will receive a single dose of CD40L-Augmented TIL. Toxicity will be evaluated at every 4 patients. The study may enroll 16-20 patients to reach 12 TIL safety evaluable patients.
  Interventions: Drug: Cyclophosphamide; Drug: Fludarabine; Drug: Interleukin-2; Drug: TIL Product
- Cohort 1: Phase II efficacy trial (Experimental): If there are 2 responders or more, the trial will continue to enroll additional 14 patients in the 2nd stage.
  Interventions: Drug: Cyclophosphamide; Drug: Fludarabine; Drug: Interleukin-2; Drug: TIL Product
- Cohort 2: Rare melanoma subtypes (Experimental): Cohort 2 will include n=10 patients with the rare melanoma histological subtypes of mucosal or uveal melanoma and will be used to assess feasibility and toxicity of the treatment in those rare melanoma subtypes.
  Interventions: Drug: Cyclophosphamide; Drug: Fludarabine; Drug: Interleukin-2; Drug: TIL Product

INTERVENTIONS:
Drug: Cyclophosphamide — Part of lymphodepletion regimen.
Drug: Fludarabine — Part of lymphodepletion regimen.
Drug: Interleukin-2 — Standard of care.
Drug: TIL Product — Tumor-infiltrating lymphocytes are an investigational, personalized adoptive cell therapy.

SUMMARY:
This is a phase I/II clinical trial of a single dose of CD40L-augmented TIL administered in patients with advanced melanoma (Cohort 1: Cutaneous acral melanoma, cutaneous non-acral melanoma, (n=26); Cohort 2: Mucosal melanoma, uveal melanoma, (n=10)). Patients will undergo an excision of a readily accessible tumor for preparation of TIL. Eligible patients with progressive disease after standard of care therapy will undergo lymphodepletion with cyclophosphamide and fludarabine followed by CD40L-augmented TIL and standard of care bolus dose interleukin-2 (short-course IL-2).

ELIGIBILITY:
Inclusion Criteria:

* Participants must have histologically confirmed, unresectable (Stage III/IV) or metastatic melanoma as follows: Cutaneous, non-acral, melanoma (including melanoma of unknown primary); Cutaneous acral melanoma; Mucosal melanoma; Ocular melanoma (including uveal, iris, conjunctival melanoma).
* Participants must have failed, be refractory to, or unable to tolerate at least one line of standard of care in the opinion of the Investigator. For participants with cutaneous non-acral melanoma, standard of care therapy includes a PD-1/L1 or combination therapy with anti-PD1 and anti-CTLA4 or combination therapy of anti-PD1 and anti-LAG3 or if BRAF V600 activating mutation positive, a BRAF ± MEK inhibitor. Participants are allowed to be enrolled in this trial if they failed one line of any of those standards of care therapy regimens.
* Any systemic therapy, including anti-cancer monoclonal antibodies, must have been completed at least 4 weeks from the start of lymphodepleting therapy, and any prior therapy-related AEs must have resolved to Grade ≤ 1 except for alopecia and vitiligo.
* Participants must be ages ≥18. Additionally, participants who are ≥ 65 years of age may need to undergo a cardiology evaluation including a cardiac stress test or coronary computed tomography after which they must be deemed to be low/acceptable risk. This cardiac evaluation may be omitted for patients who underwent testing within 6 months and have no interval change in cardiopulmonary clinical status. Note 1: Cardiac stress test may be omitted for patients ≥65 years old (y/o) who are fully functional with no relevant medical comorbidities and are able to carry ≥4 METS activities at baseline. For patients who demonstrate abnormal cardiac stress test cardiac evaluation by cardiologist will be done and if deemed low acceptable risk, will be allowed to participate in this trial per PI discretion. Cardiac stress test may be indicated for any patient <65 y/o who have relevant medical comorbidities or demonstrate clinically worrisome symptoms. Note 2: While age preference will be between 18-75 years, this study allows age >75 years if the patient meets eligibility criteria and demonstrates no significant medical comorbidities per PI.
* ECOG performance status of 0 or 1.
* Participants must have adequate organ and marrow function as defined within the protocol.
* Seronegative for Human immunodeficiency virus (HIV) antibody, hepatitis B surface antigen, and hepatitis C (HCV) antibody (if HCV antibody positive, must be tested for HCV RNA, which must be negative to be eligible).
* Participants with brain metastases are eligible provided that the brain metastases have been successfully treated with stereotactic radiosurgery or resection and clinically stable for at least 4 weeks (±14 days). Note: Participants who develop brain metastases after tumor harvest and/or lymphodepleting therapy will be allowed to remain on study and may proceed with cell therapy after undergoing definitive radiation therapy and/or surgery. For those participants who develop brain metastases during lymphodepleting therapy and undergo definitive radiation therapy and/or surgery careful decision will be made to proceed with TIL infusion after discussion with treating physician, neurosurgeon, radiation oncologist and PI.
* Women of child-bearing potential must have a negative pregnancy test.
* The effects of CD40L-augmented TIL on the developing human fetus are unknown. For this reason and because TIL agents, as well as other therapeutic agents used in this trial including IL-2 are known to be teratogenic, both males and females of childbearing potential must be willing to practice birth control starting with screening through 1 year after the last study drug is administered for females or 6 months for males.
* Should a woman become pregnant or suspect she is pregnant while she or her partner are participating in this study, she should inform her treating physician immediately.
* Ability to understand and the willingness to sign a written informed consent document.
* Participants should have at least one surgically accessible lesion for tumor harvest for preparation of TIL, and at least one RECIST v1.1 measurable lesion after tumor harvest to follow for response assessment. Note: Tumor harvest lesion will be considered as target lesion if after harvest remaining portion of tumor meets RECIST v1.1 measurable lesion criteria.

Exclusion Criteria:

* Participants, regardless of age, who have a current or past medical history of ischemic heart disease, or clinically significant atrial or ventricular rhythm abnormality are excluded unless they undergo a cardiac stress test and cardiology clearance examination and are determined to be low or acceptable risk.
* Participants with either a primary immunodeficiency disorder (i.e., severe combined immunodeficiency syndrome) or acquired immunodeficiency disorders (such as HIV/AIDS).
* Pregnant women are excluded from this study because the agents used in this study have teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with CD40L-augmented TIL or the other agents in the study, breastfeeding should be discontinued if the mother is enrolled in the study.
* Participants taking systemic steroid therapy (other than replacement therapy or prednisone equivalent of ≤10mg daily) or therapy with any immunosuppressive medications such as mycophenolate mofetil (MMF). Participants who require more than 10mg of prednisone or equivalent other steroid therapy should taper their steroid therapy to 10 mg prednisone 1 week prior to planned first interventional drug therapy (lymphodepleting therapy). Participants who are on baseline replacement therapy or prednisone equivalent of ≤10mg daily and require stress doses of steroid therapy will be allowed to receive stress dose steroids during the trial interventions. Participants who require dapsone for pneumocystis pneumonia (PCP) prophylaxis during TIL therapy are eligible.
* Participants who have a history of severe immediate hypersensitivity reaction to the study agents including cyclophosphamide, fludarabine, or IL-2 or any of their constituents.
* Participants with a left ventricular ejection fraction (LVEF) ≤ 45% or New York Heart Association (NYHA) functional classification > 1.
* Forced expiratory volume (FEV1) ≤ 60% of predicted value and DLCO (corrected) < 60% of predicted value. Participants who underwent pulmonary function testing within 6 months of screening may omit PFTs if they demonstrate stable cardiopulmonary status.
* Participants who, in the opinion of the Investigator, have a medical condition that would subject the patient to prohibitive risk by participation in this study, or who may be unable to safely complete tumor harvest, lymphodepletion regimen, TIL infusion, or aldesleukin administration.
* Participants with active infections requiring antibiotics.
* Participants with active autoimmune diseases currently requiring systemic treatment with immunosuppressive doses of corticosteroids (>10 mg of prednisone-equivalent daily dosing), immunosuppressive biologic agents, or disease modifying antirheumatic drug agents (DMARDs).
* Patients who received prior live cell therapy are excluded, unless express written permission is provided by the clinical PI.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2029-05 (Estimated); Study Completion 2030-05 (Estimated)

PRIMARY OUTCOMES:
Phase I: Treatment Emergent Adverse Events (TEAE) | Up to 28 days post TIL
  The proportion of patients who experience a TEAE
Phase II: Objective Response Rate | Up to 60 Months
  The proportion of response evaluable patients.

SECONDARY OUTCOMES:
Duration of response | Up to 60 Months
  Duration of response (DOR) in months, of the total response-evaluable patients.
Progression Free Survival (PFS) | Up to 60 Months
  Progression Free Survival (PFS) in months of the total safety-evaluable patients, and the total treated patients.
Overall survival | Up to 60 Months
  Overall Survival (OS) in months of the total safety-evaluable patients, and the total treated patients.

CONTACTS AND LOCATIONS:
Overall Officials: Lilit Karapetyan, MD, Principal Investigator — Moffitt Cancer Center
Locations (1):
- Moffitt Cancer Center, Tampa, Florida, United States